CLINICAL TRIAL: NCT03723746
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Day Dose Study to Assess the Safety and Tolerability of JNJ-67670187 in Healthy Participants
Brief Title: A Study to Evaluate the Safety and Tolerability of JNJ-67670187 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108532; 2018-002287-81 (EudraCT Number); 67670187IBD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1: Dose 1 or Placebo (Part 1 - SD) (Experimental): Participants will receive a single oral dose (single day [SD] Dose 1) of either JNJ-67670187 or placebo capsules after an overnight fast on Day 1 of Part 1.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 2: Dose 2 or Placebo (Part 1 - SD) (Experimental): Participants will receive a single oral dose (Dose 2) of either JNJ-67670187 or placebo capsules after an overnight fast on Day 1 of Part 1.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 3: Dose 1 or Placebo (Part 2 - MD) (Experimental): Participants will receive an oral dose (Multiple Day [MD] Dose 1) of either JNJ-67670187 or placebo capsules once daily for 14 days without antibiotic pretreatment after an overnight fast in Part 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 4:Antibiotic + Dose 1 or Placebo (Part 2 - MD) (Experimental): Participants will receive pretreatment with an oral antibiotic, followed by an oral dose (Dose 1) of either JNJ-67670187 or placebo capsules once daily for 14 days after an overnight fast in Part 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 5: Dose 2 or Placebo (Part 2 - MD) (Experimental): Participants will receive an oral dose (Dose 2) of either JNJ-67670187 or placebo capsules once daily without antibiotic pretreatment for 14 days after an overnight fast in Part 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 6:Antibiotic + Dose 2 or Placebo (Part 2 - MD) (Experimental): Participants will receive pretreatment with an oral antibiotic, followed by an oral dose (Dose 2) of either JNJ-67670187 or placebo capsules once daily for 14 days after an overnight fast in Part 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 7 (Optional): Laxative + Dose 2 or Placebo (Part 3) (Experimental): Participants may receive pretreatment with an oral laxative, followed by an oral dose (Dose 2) of either JNJ-67670187 or placebo capsules once daily for 14 days after an overnight fast in Part 2. Cohort 7 (Part 3) will only be conducted if the strains are not detected in microbial analysis of Parts 1 and 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 8 (Optional):Antibiotic+Laxative+Dose 2/Placebo(Part 3) (Experimental): Participants may receive pretreatment with an oral antibiotic and oral laxative, followed by an oral dose (Dose 2) of either JNJ-67670187 or placebo capsules once daily for 14 days after an overnight fast in Part 2. Cohort 8 (Part 3) will only be conducted if the strains are not detected in microbial analysis of Parts 1 and 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo
- Cohort 9 (Optional): Dose 2 or Placebo (Part 3) + Biopsy (Experimental): Participants may receive an oral dose (Dose 2) of either JNJ-67670187 or placebo capsules once daily for 14 days after an overnight fast in Part 2. After final dosing collection of sigmoid biopsies will be performed. Cohort 9 (Part 3) will only be conducted if the strains are not detected in microbial analysis of Parts 1 and 2.
  Interventions: Biological: JNJ-67670187; Biological: Placebo

INTERVENTIONS:
Biological: JNJ-67670187 — Participants in Cohorts 1, 3 and 4 will receive Dose 1 and participants in Cohorts 2, 5, 6, 7, 8 and 9 will receive Dose 2.
Biological: Placebo — Participants will receive matching placebo in all cohorts.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single and multiple day dose of JNJ-67670187 compared to placebo.

DETAILED DESCRIPTION:
This study will be a Phase 1 randomized double-blind, placebo controlled multi dose study in up to 144 adult healthy volunteers. The safety, tolerability and impact on the microbiome following intake of oral dose of JNJ-67670187 for up to 14 days will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) inclusive, and a body weight of at least 50 kilogram (kg)
* Be otherwise healthy on the basis of physical examination, medical history, and vital signs, and 12 lead electrocardiogram (ECG) performed at screening and at admission
* Be otherwise healthy on the basis of clinical laboratory tests performed at screening and at admission. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant
* All women of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on day of admission
* Must have normal bowel movements

Exclusion Criteria:

* Has a positive serum pregnancy test at screening, a positive urine pregnancy test, or is a female still lactating prior to study intervention administration
* An active cigarette smoker or has quit cigarette smoking within the previous 6 months
* Has a positive urine toxicology screen at screening or at admission for substances of abuse including but not limited to cocaine, cannabinoids, amphetamines, benzodiazepines, barbiturates, opiates, tricyclic antidepressants and methadone
* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal (GI) disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Has an active systemic or GI acute or chronic infection as determined by appropriate clinical screening and laboratory tests

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Part 1 Single Day (SD) Dose: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events as a Measure of Safety and Tolerability | 3 Months post final dose or up to Day 84
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are AEs which will occur between administration of study drug and 3 months or up to Day 84 that were absent before treatment or that worsened relative to pre-treatment state. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 2 Multiple Day (MD) Dose : Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events as a Measure of Safety and Tolerability | 3 Months post final dose or up to Day 98
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are AEs which will occur between administration of study drug and 3 months or up to Day 98 that were absent before treatment or that worsened relative to pre-treatment state. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 1 SD: Number of Participants With Abnormalities in Vital Signs, Physical Examinations, Electrocardiogram (ECG), and Clinically Significant Laboratory Findings as a Measure of Safety and Tolerability | Predose up to Day 84
  Number of participants with abnormalities in vital signs, physical examinations, ECG and clinically significant laboratory findings will be reported.
Part 2 MD: Number of Participants With Abnormalities in Vital Signs, Physical Examinations, Electrocardiogram (ECG), and Clinically Significant Laboratory Findings as a Measure of Safety and Tolerability | Predose up to Day 98
  Number of participants with abnormalities in vital signs, physical examinations, ECG and clinically significant laboratory findings will be reported.

SECONDARY OUTCOMES:
Detection and Abundance of JNJ-67670187 | Pre-dose, up to Day 82 (SD) and up to Day 98 (MD)
  Stool assessment will be done to characterize the presence of JNJ-67670187.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Clinical Pharmacology Unit, Merksem, Belgium
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands